CLINICAL TRIAL: NCT02992977
Title: A Phase 1 Study of Safety and Tolerability of AutoSynVax™ Vaccine as a Single Agent in Subjects With Advanced Cancer
Brief Title: Safety and Tolerability Study of AutoSynVax™ Vaccine in Subjects With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: To enable development of an enhanced version of the vaccine.
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-600-01
Record Dates: First submitted 2016-12-09; First posted 2016-12-14 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Advanced Cancer
Keywords: Vaccine, neoantigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AutoSynVax™ vaccine (Experimental): AutoSynVax™ vaccine + QS-21 Stimulon® adjuvant
  Interventions: Biological: AutoSynVax™ vaccine

INTERVENTIONS:
Biological: AutoSynVax™ vaccine — AutoSynVax™ vaccine + QS-21 Stimulon® adjuvant

SUMMARY:
Open-label Phase 1 study of AutoSynVax™ vaccine with QS-21 Stimulon® adjuvant in subjects with advanced cancer

DETAILED DESCRIPTION:
This is an open-label Phase 1 study to determine the safety and tolerability of single-agent treatment with AutoSynVax™ vaccine with QS-21 Stimulon® adjuvant in subjects with advanced cancer that is refractory to standard therapies and a life expectancy of ≥6 months from the time tissue is obtained. A minimum of 6 (≤20) subjects will be enrolled to receive every other week subcutaneous injection of 240 μg AutoSynVax™ vaccine + 50 μg QS-21 Stimulon® adjuvant for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

Prior to vaccine production -

1. Diagnosis of advanced cancer (solid tumor) that:

   1. May be receiving or about to start another line of therapy.
   2. If on a line of therapy or about to start a new line of therapy, it is anticipated that the treatment may provide short-term tumor control.
2. Available tissue from an archival tissue sample or tissue from a biopsy done during the initial screen, or both. If archival tissue is not available or tissue is not mainly tumor, subjects must be willing to undergo a biopsy or surgery to remove some or all of their tumor for next generation sequencing. New tissue should be obtained prior to starting a new line of therapy, if applicable.
3. Minimum estimated life expectancy of 6 months.
4. Age 18 years or older.
5. Signed written informed consent to allow transfer of tumor tissue and production of vaccine.
6. Discussion about each patient should occur with the Medical Monitor to confirm eligibility.

Prior to Treatment -

Patients who had vaccine manufactured but were treated with an additional line of treatment may start vaccine if they continue to meet the remaining eligibility criteria.:

1. Diagnosis of advanced cancer (solid tumor) that is refractory to standard therapies.
2. Signed written informed consent for treatment.
3. Minimum estimated life expectancy of 3 months.
4. Eastern Cooperative Oncology Group (ECOG) performance status <2.
5. Adequate bone marrow function (absolute neutrophil count [ANC] ≥1,500/mm^3; absolute lymphocyte count [ALC] ≥500/mm^3; platelet count 100,000/mm^3), adequate liver function (serum glutamic oxaloacetic transaminase [SGOT]/aspartate aminotransferase [AST] and alkaline phosphatase <2.5 times the institutional upper limit of normal [IULN], total bilirubin <1.5 mg/dL), and adequate renal function (creatinine <1.5 x IULN).
6. Adequate cardiac function (New York Heart Association [NYHA] class ≤II).
7. All participants (males and females) must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study treatment and for the duration of study participation.

Female subjects of childbearing potential should have a negative serum pregnancy test at pre-treatment visit and within 72 hours prior to receiving the first dose of study medication.

Female subjects of childbearing potential must agree to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity prior to receiving the first dose of study medication through 30 days after the last dose of study medication.

Exclusion Criteria:

Subjects must not meet any of the following exclusion criteria at the time of tumor procurement. All exclusion criteria must be confirmed prior to treatment.

1. Diagnosis of immunodeficiency or actively receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
2. Corticosteroid dependency.
3. Requirement for immunosuppressive medication aside from corticosteroids.
4. Active or history of any autoimmune disease (subjects with diabetes type 1, vitiligo, psoriasis, hypo-, or hyperthyroid disease not requiring immunosuppressive treatment are eligible) or immunodeficiencies.
5. History of treated or untreated brain metastases or leptomeningeal spread of disease.
6. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
7. Known medical, psychiatric or substance abuse disorders that would preclude participation in the study.
8. Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Known to be positive for human immunodeficiency virus (HIV). Testing is not required in the absence of history or high index of suspicion.
10. Intolerance of prior immunotherapy treatment necessitating cessation of therapy.
11. History of intolerance or allergic reactions attributed to compounds of similar chemical or biologic composition to AutoSynVax™ vaccine or QS-21.
12. Women who are pregnant or breastfeeding.
13. Inability to comply with protocol.

Prior to Treatment - Subjects must not meet any of the following exclusion criteria prior to treatment in addition to the other exclusion criteria listed above.

1. Receipt of anticancer medications or investigational drugs within the following intervals before first administration of study drug:

   1. ≤14 days for chemotherapy, targeted small molecule therapy, anticancer hormone therapy or radiation therapy. Subjects must also not have had radiation pneumonitis as a result of treatment, and cannot participate in the study if they are on chronic corticosteroids for radiation pneumonitis or other reasons. A 1-week washout is permitted for palliative radiation to non-CNS disease with sponsor approval.
   2. Note: Bisphosphonates and denosumab are permitted medications. Novel imaging agents that have Phase 1 safety data and have not demonstrated therapeutic activity are also permitted.
   3. ≤28 days for a prior immunotherapy.
   4. ≤28 days for prior monoclonal antibody used for anticancer therapy with the exception of denosumab.
   5. ≤7 days for immunosuppressive-based treatment for any reason. Systemic corticosteroids are not allowed.

      Note: Use of inhaled or topical corticosteroid use for radiographic procedures is permitted.

      Note: Patients receiving physiologic steroid replacement for adrenal insufficiency are eligible (i.e. < 10 mg prednisone per day).

      Note: The use of physiologic corticosteroid replacement therapy may be approved after consultation with the sponsor.
   6. ≤28 days before the first dose for all other investigational study drugs or devices.
2. Receipt of other investigational agents or other anticancer therapies during treatment with AutoSynVax™ vaccine.
3. Receipt of a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergence Adverse Events (Safety and Tolerability) | From first administration to 30 days from last dose.
  AEs, irAEs, according to NCI CTCAE version 4.03.
Recommended dose for further development | 28 days from first dose
  After 2 doses (administered every 2 weeks), if there are <2 treatment-limiting toxicities (TLTs) in the first 6 subjects, AutoSynVax™ vaccine will be considered safe for further development.

SECONDARY OUTCOMES:
Overall survival (OS) | From first administration until death, or up to study duration (18 - 24 months)
  Duration of survival
Progression-free survival (PFS) | 6 Months after last dose is administered.
  From time of first administration per RECIST v1.1
Objective response rate (ORR) | 6 Months after last dose is administered.
  From time of first administration per RECIST v1.1
T-cell response | 6 Months after last administration.
  T-cell response to tumor specific neo-epitopes in the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (2):
- United States (2):
  - School of Medicine at the University of Miami, Miami, Florida
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No